CLINICAL TRIAL: NCT03585842
Title: French Validation of the Dual Diagnosis Screening Interview (F_DDSI)
Acronym: F_DDSI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-396; 2017-A03042-51 (Other: 2017-A03042-51)
Record Dates: First submitted 2018-06-28; First posted 2018-07-13 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-06

CONDITIONS: Substance Related Disorders; Psychiatric Comorbidities
Keywords: Scale Translation; Substance Use Disorder; Comorbidities psychiatric
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-test group: Patients from CMP B coming for consultation or day hospital
  Interventions: Other: No intervention
- Test group: Patients suffering from DSMV substance use disorder with one or more psychiatric comorbidities
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
In France, there are no tools for screening psychiatric comorbidities for individuals with Substance Use Disorders. The literature shows that the cooccurrence of these psychiatric disorders in the same individual is frequent. It negatively impacts the healing prognosis, complicates the diagnostic processes and the type of care to be introduced for patients. The creation of reliable, fast and easy-to-use tools for caregivers and researchers is therefore necessary to improve quantitatively and qualitatively the care of patients. There is a Spanish scale that meets these criteria, the Dual Diagnostic Screening Interview (S_DDSI). The main objective of this study is to validate the DDSI in French. The secondary objectives are the evaluation of the psychometric qualities of F_DDSI (French version) and adaptation of this scale into an application for Android and iOS.

DETAILED DESCRIPTION:
Type of study: Cross-sectional exploratory, non-interventional Research category : research involving the human person, category III Number of centers: 2 French centers in Auvergne region Study Performance

The methodology includes 3 phases :

Phase 1: translations / back-translation / expert consensus, comes in four stages.

A) The translation of the Spanish scale (LO) will be carried out by different translators into two distinct French versions (LC1 and LC2).

B) These two versions will then be compared by a consensus of experts to lead to the first version of the scale in French (V1-LC) C) Which will then be translated back into Spanish (B-LC1). D) This last version will itself be compared with the S_DDSI to retain or reject items, instructions or response format too discordant that will have to be modified by consensus on proposal of the experts or go back through the previous stages of the translation. The expert consensus involved in steps B) and D) will apply the DELPHI method to accept, reject or re-evaluate each of the items.

Phase 2: Pre-test Pre-testing the scale, through individual interviews with a dozen patients, in order to measure the reactions and the degree of comprehension of the instructions, the items and the clarity of the response format. Items assessed as unclear by at least 2 patients will need to be reassessed. The experts will then have to provide new proposals which will in turn have to be reevaluated by the patients.

Phase 3 : Scale Test The test of the scale obtained, will be conducted with 200 patients through individual interviews. The results obtained will make it possible to test the acceptability of the questionnaire by analyzing the response rate for each items and measure the psychometric qualities of the tool (validity of the internal structure, multi-dimensionality, internal coherence of each sub-dimension). The Gold Standard used for this last phase is the MINI.

Patients Phase 2: Subjects participating in the pre-test phase will only be recruited from the CMP B patients coming for consultation or day hospital.

Phase 3: For the test phase of the scale, the subjects must be patients suffering from DSMV substance use disorder with one or more psychiatric comorbidities.

In phase 2 and 3, the inclusion time of the subjects corresponds to the filling time of the scales.

ELIGIBILITY:
Inclusion Criteria:

Phase 2 : Patients coming for consultation in the department or day hospital Phase 3: Subjects presenting for one or more substances a diagnosis of Substance Use Disorders (SUD) according to the DSMV criteria.

Exclusion Criteria:

Phase 2

* Subject who do not understand French
* Subject unable to answer questions cognitively

Phase 3

* Subject who do not understand French
* Subject unable to answer questions cognitively
* Subjects with a mental disorder of the axis I of the DSMIV not stabilized making impossible the filling of the questionnaire (in particular acute states delusional and dissociative)
* Subjects who participated in the pre-test phase (2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Both female and male participants of 18 years old and more are being studied.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2018-03-14 (Actual); Primary Completion 2019-01-31 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
The response rates for each of the item composing the instrument | From March 14, 2017 to June 2019
Psychometric qualities of the new scale | From March 14, 2017 to June 2019
  Sensitivity, specificity, and the positive and negative predictive values for each disorder measured by the DDSI will be calculated in comparison with the MINI

CONTACTS AND LOCATIONS:
Overall Officials: Georges BROUSSE, PhD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (2):
- France (2):
  - CHU de Clermont-Ferrand, Clermont-Ferrand, Auvergne
  - CH Etienne Clémentel, Enval, Auvergne